CLINICAL TRIAL: NCT05385107
Title: Value of PCT When Diagnosing Candidemia
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, Associate Profesor, Senior Consultant, Karolinska University Hospital
Other Study IDs: EPN 2017/806-31 (Candida-PCT)
Record Dates: First submitted 2021-12-12; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: The Value of Procalcitonin in Patients With Suspected Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum procalcitonin concentration

SUMMARY:
This study is a retrospective analysis to identify and compare the shift in inflammatory biomarkers in ICU patients immediately before and after the first identification of candidemia.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria (all has to be fullfilled):

* ICU patients with blood cultures showing growth of Candida species
* clinical records including daily data on WBC, CRP, Procalcitonin and body temperature

Exclusion Criteria:

* Age lower than 18 years
* blood cultures with growth of Candida species before ICU admission
* incomplete records of daily WBC, CRP, Procalcitonin or body temperature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Absolute procalcitonin concentration | 9 days
Shift (trend) procalcitonin concentration | 9 days

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
No plan